CLINICAL TRIAL: NCT05508204
Title: BION-1301 - A Phase 1, Open-label, Single Subcutaneous Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Japanese Healthy Subjects
Brief Title: Open-label Safety and PK Study of BION-1301 in Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHK02-01
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: Open-label, single ascending dose study in Japanese healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): A single dose of BION-1301 will be administered subcutaneously on Day 1 at dose level A
  Interventions: Drug: BION-1301
- Cohort B (Experimental): A single dose of BION-1301 will be administered subcutaneously on Day 1 at dose level B
  Interventions: Drug: BION-1301
- Cohort C (Experimental): A single dose of BION-1301 will be administered subcutaneously on Day 1 at dose level C
  Interventions: Drug: BION-1301

INTERVENTIONS:
Drug: BION-1301 — A solution for SC injection administered as a single dose

SUMMARY:
Phase 1, open-label study designed to evaluate safety, tolerability, pharmacokinetic, and pharmacodynamic of multiple doses of BION-1301 in Japanese healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1 study of BION-1301, a first-in-class humanized IgG4 anti-a proliferation-inducing ligand (APRIL) monoclonal antibody. This is a single-center, open-label study designed to evaluate safety, tolerability, pharmacokinetic, and pharmacodynamic of a single subcutaneous dose of BION-1301 in Japanese healthy subjects in 3 dose level cohorts. The study will enroll up to 36 Japanese subjects across 3 dose level cohorts.

ELIGIBILITY:
Inclusion Criteria:

* First generation Japanese (confirmed at screening). The definition of first generation is the subject, the subject's biological parents, and the subject's biological grandparents are of exclusively Japanese origin and were born in Japan.
* Body mass index (BMI) between 18 and 30 kg/m^2, inclusive, at screening with a weight of at least 47 kg.
* In good health, as determined by medical history, physical examination, vital signs assessment, 12-lead ECG, and clinical laboratory evaluations within normal reference ranges or outside of normal reference ranges considered not clinically relevant by the investigator
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test, must agree to try to not become pregnant, must agree to consistently use highly effective contraceptive methods, and must agree not to breastfeed or donate ova for a period as defined in the study protocol.
* Male subjects must agree to use highly effective contraceptive methods and must not donate sperm for a period as defined in the study protocol.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of malignancy during the last 3 years; exceptions include adequately treated basal cell carcinoma and squamous cell carcinoma of the skin
* Confirmed systolic blood pressure >140 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, and pulse rate >100 or <40 beats per minute at either screening or predose on Day 1.
* Received a live (attenuated) vaccine(s) within 3 months prior to check-in and/or a vaccine(s) that do not contain live microorganism(s) within 14 days prior to check-in.
* Have previously completed or withdrawn from this study or any other study investigating BION-1301, and have previously received BION-1301.
* Positive urine drug screen, alcohol test, or cotinine test at screening or check-in.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BION-1301 | Day 85
  Number of subjects with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs); changes from baseline in safety parameters; and number of subjects with injection site reactions

SECONDARY OUTCOMES:
Pharmacokinetics-Cmax | Day 85
  Maximum plasma concentration
Pharmacokinetics-Tmax | Day 85
  Time at which the maximum plasma concentration (Cmax) occurs
Pharmacokinetics-AUC∞ | Day 85
  Area under the plasma concentration-time curve from dosing (time zero) extrapolated to infinity
Pharmacokinetics-AUClast | Day 85
  Area under the plasma concentration-time curve from dosing (time zero) to the time of the last measured concentration
Pharmacokinetics-t1/2 | Day 85
  Time required for the drug concentration to decrease by a factor of one-half in the terminal phase
Pharmacokinetics-CL/F | Day 85
  Serum concentration after single dose will be measured and the apparent oral clearance will be calculated
Pharmacokinetics-Vz/F | Day 85
  Serum concentration after single dose will be measured and the apparent volume of distribution will be calculated
The effect of BION-1301 on pharmacodynamic (PD) parameters | Day 85
  Changes in immunoglobulin levels (IgA, IgG, and IgM)
The levels of anti-drug antibodies | Day 85
  Blood anti-drug antibodies (ADA) and neutralizing antibody (NAb) levels

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Jones-Burton, M.D., Study Director — Chinook Therapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Research, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No